CLINICAL TRIAL: NCT07232797
Title: Clinical Evaluation of Pit and Fissure Sealants Placed by Intern Dental Students After Tele-demonstration Technique
Brief Title: Sealant Application by Interns After Tele-demonstration
Acronym: TESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, ahmed elsebaai, lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DU:0240221004
Record Dates: First submitted 2025-09-20; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Dental Caries; Prevention; Education
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: parallel assignment with split mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tele-demonstration group (Experimental): trained via pre-recorded video
  Interventions: Behavioral: traditional demonstration group
- traditional demonstration group (Active Comparator): trained via in person clinical demo
  Interventions: Behavioral: tele-demonstration

INTERVENTIONS:
Behavioral: tele-demonstration — tele-education via pre-recorded video tutorial for sealant application
  Arms: traditional demonstration group
Behavioral: traditional demonstration group — direct in person clinical demonstration of sealant application
  Arms: tele-demonstration group

SUMMARY:
Abstract

Background:

Dental caries remains a major public health issue worldwide, particularly among children. Pit and fissure sealants represent a high-quality, evidence-based preventive measure. However, ensuring the reliability of their application by newly graduated intern dental students trained through tele-education remains an emerging area of growing interest.

Objective:

To evaluate the clinical success rate of pit and fissure sealants placed by intern dental students following tele-demonstration training versus traditional training approaches.

Methods:

This randomized controlled trial involved 100 mandibular first permanent molars in 50 children aged 7 to 9 years, treated by 20 dental interns assigned to two groups using a split-mouth design. One group received direct clinical demonstration, while the other received tele-education via a pre-recorded video. Sealant retention and marginal discoloration were assessed after a 3-month period.

Keywords:

tele-dentistry, tele-demonstration, tele-education, intern dental students, sealants, first permanent molar

DETAILED DESCRIPTION:
Abstract

Background:

Dental caries continues to be one of the most prevalent chronic diseases worldwide, with the highest incidence occurring among school-aged children. The occlusal surfaces of permanent molars are particularly susceptible due to their deep pits and fissures, which favor plaque accumulation and limit effective cleaning. The application of pit and fissure sealants has been widely recognized as an evidence-based preventive strategy that provides a physical barrier against cariogenic challenges. The quality and longevity of sealant placement, however, largely depend on the clinician's skill and adherence to proper clinical protocols. In recent years, the integration of tele-dentistry into dental education-specifically through tele-demonstration and tele-education-has gained growing attention as a means to enhance learning accessibility, particularly during times of restricted clinical training opportunities. Nevertheless, the clinical efficacy of procedures performed by newly graduated intern dental students following such digital training remains insufficiently explored.

Objective:

This study aimed to evaluate and compare the clinical performance and success rate of pit and fissure sealants applied by intern dental students trained through a tele-demonstration video-based module versus those trained through traditional chair side (face-to-face) demonstration. The primary endpoint was sealant retention, while secondary outcomes included marginal discoloration after a 3-month follow-up period.

Methods:

A randomized controlled split-mouth clinical trial was conducted on a total of 100 mandibular first permanent molars in 50 healthy children aged 7-9 years attending the pediatric dental clinics. Twenty dental interns participated in the study and were randomly allocated into two equal groups based on the mode of training received. Group A interns received conventional in-person clinical demonstrations of the sealant application procedure by a pediatric dentistry specialist. Group B interns received remote tele-demonstration training via a standardized pre-recorded instructional video detailing each clinical step, from tooth isolation and acid etching to sealant application and curing. Clinical evaluation of sealant retention and marginal discoloration after 3 months period. Data were statistically analyzed and p value significance set at p < 0.05.

Keywords:

tele-dentistry, tele-demonstration, tele-education, dental interns, pit and fissure sealants, preventive dentistry, first permanent molar

ELIGIBILITY:
Inclusion Criteria:

* Children age extending from 7 - 9 years
* bilaterally caries-prone, sound lower first permanent molars

Exclusion Criteria:

* Teeth with initial carious lesions or cavitated lesions
* children parents or legal guardians were unable to provide informed consent.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
sealant retention | 3 months post application
  The retention rate of sealants was evaluated according to 'Simonsen's criteria' [10]: (a) Total retention - complete coverage of the occlusal surface by the sealant (score 0); (b) Partial loss - sealant present with visible fractures or partial loss of material (score 1); and (c) Total loss - complete absence of the sealant from the occlusal surface (score 2).

SECONDARY OUTCOMES:
marginal discoloration | 3 months post application
  Marginal discoloration was also assessed as either present or absent, as its presence may indicate early signs of marginal leakage.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-sebaai, Lecturer, Principal Investigator — Faculty of dentistry, Delta University, Egypt
Locations (1):
- Operative Dentistry Department, Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Raw data could be shared
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publishing
Access Criteria: Principal investigator email